CLINICAL TRIAL: NCT03811158
Title: The Diaphragm Activity Level and Cardiopulmonary Function Between Heated Humidified High-Flow Nasal Cannula and Unheated Humidified High-Flow Oxygen Mask in Acute Exacerbation of COPD Patients as Post-Extubation Respiratory Support
Brief Title: The Edi Level and Cardiopulmonary Function Between HHHFNC and Unheated Humidified High-Flow Oxygen Mask in COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult to recruit participants
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PL-201705001-M
Record Dates: First submitted 2019-01-14; First posted 2019-01-22 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Chronic Obstructive Lung Disease; Respiratory Insufficiency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patents with COPD exacerbation who were intubated for respiratory failure will all enrolled to this study. Participants will be studied on 2 consecutive days and random assigned with crossover. The primary outcome measure is the diaphragm electrical activity. The secondary outcome measures include the cardiopulmonary function, length of hospital stay, and re-intubation rate.
Who Masked: Investigator
Masking Description: All data will be decoded before biostatics analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HHHFNC group (Experimental): On HHHFNC FiO2 will setting as same as SBT before extubation Flow rate: 50L/min
  Interventions: Device: HHHFNC
- UHFOM group (Sham Comparator): On Aerosol mask FiO2 will setting as same as SBT before extubation Flow rate: 15L/min
  Interventions: Device: UHFOM

INTERVENTIONS:
Device: HHHFNC — Prospective, randomized crossover control trial, single ICU. Patents with COPD exacerbation who were intubated for respiratory failure will all enrolled to this study. Participants will be studied on 2 consecutive days and random assigned with crossover.
  Other Names: Study group
  Arms: HHHFNC group
Device: UHFOM — Prospective, randomized crossover control trial, single ICU. Patents with COPD exacerbation who were intubated for respiratory failure will all enrolled to this study. Participants will be studied on 2 consecutive days and random assigned with crossover.
  Other Names: Control group
  Arms: UHFOM group

SUMMARY:
Patients with COPD exacerbation usually need respiratory support after extubation. Recently, HHHFNC has been used in both adult and neonates with post-extubation respiratory support. Studies indicate that HHHFNC has seminar efficacy compared to non-invasive positive pressure ventilation and superior than conventional oxygen therapy. There are no clinical data of diaphragm electrical activity and cardiopulmonary function for using HHHFNC and UHFOM as post-extubation respiratory support.

DETAILED DESCRIPTION:
Objectives： The aim of this study is to compare the Edi level and cardiopulmonary parameters between heated humidified high-flow nasal cannula (HHHFNC) versus unheated high-flow oxygen mask (UHFOM) in acute exacerbation of chronic obstructive pulmonary disease (COPD) patients with post-extubation respiratory support. This is the first clinical trial to investigate and analysis the variations of cardiopulmonary parameters and Edi level between HHHFNC and UHFOM in adult patients.

ELIGIBILITY:
Inclusion Criteria:

1. AE of COPD received intubation and ready to be weaning
2. P/F ratio > 200 during SBT before extubation

Exclusion Criteria:

1. Unable to insert NG tube
2. Refuse to re-intubated when respiratory failure after extubation
3. Planned NIV use after extubation
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Diaphragm electrical activity | 2 days
  In voltage

SECONDARY OUTCOMES:
PtcO2 & PtcCO2 | 2 days
  In mmHg
Re-intubation rate | 2 days
  In %
Cardiac index | 2 days
  In L/min/m2
Hospital stay | through study completion, an average 3 months
  In days
ICU stay | through study completion, an average 1 months
  In days

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, M.Sc, Principal Investigator — ck_qq@hotmail.com
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brotfain E, Zlotnik A, Schwartz A, Frenkel A, Koyfman L, Gruenbaum SE, Klein M. Comparison of the effectiveness of high flow nasal oxygen cannula vs. standard non-rebreather oxygen face mask in post-extubation intensive care unit patients. Isr Med Assoc J. 2014 Nov;16(11):718-22. PMID 25558703
- [Result] Stephan F, Barrucand B, Petit P, Rezaiguia-Delclaux S, Medard A, Delannoy B, Cosserant B, Flicoteaux G, Imbert A, Pilorge C, Berard L; BiPOP Study Group. High-Flow Nasal Oxygen vs Noninvasive Positive Airway Pressure in Hypoxemic Patients After Cardiothoracic Surgery: A Randomized Clinical Trial. JAMA. 2015 Jun 16;313(23):2331-9. doi: 10.1001/jama.2015.5213. PMID 25980660
- [Result] Futier E, Paugam-Burtz C, Godet T, Khoy-Ear L, Rozencwajg S, Delay JM, Verzilli D, Dupuis J, Chanques G, Bazin JE, Constantin JM, Pereira B, Jaber S; OPERA study investigators. Effect of early postextubation high-flow nasal cannula vs conventional oxygen therapy on hypoxaemia in patients after major abdominal surgery: a French multicentre randomised controlled trial (OPERA). Intensive Care Med. 2016 Dec;42(12):1888-1898. doi: 10.1007/s00134-016-4594-y. Epub 2016 Oct 22. PMID 27771739